CLINICAL TRIAL: NCT06423950
Title: Feasibility of Generating Novel Translational and Therapeutic Strategies Based on a Multicenter, Pediatric and AYA Evolutionary Tumor Board (pedsETB)
Brief Title: Generating Novel Translational and Therapeutic Strategies Based on a Multicenter, Pediatric and AYA Evolutionary Tumor Board (pedsETB)
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22170
Record Dates: First submitted 2024-05-09; First posted 2024-05-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood collected at study enrollment and subsequently at designated time points:
  Screening/Baseline/Enrollment, first post pedsETB Visit, and every 12 weeks (+/- 6 weeks) or upon changes in disease status, therapeutic intervention, and/or events of special interest at the discretion of the treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Reviewed by ETB: Participants clinical history, available therapeutic options, and outcome expectations will be presented to the Evolutionary Tumor Board (ETB) along with images and pathology. Strategies and models will be presented regarding additional evolutionary ideas that can be applied.
  These ideas will be characterized (e.g. first strike-second strike, adaptive, novel sequential therapy, novel combination, novel dosing schedule, etc.).
  Interventions: Other: Peds Evolutionary Tumor Board (pedsETB)

INTERVENTIONS:
Other: Peds Evolutionary Tumor Board (pedsETB) — The pedsETB consists of evolutionary biologists, mathematicians, research scientists, statisticians, data scientists, radiologists, pathologists, oncologists (surgical, radiation, medical, and pediatric), and clinical trial coordinators. The pedsETB membership is inclusive of members from the participating institutions. The pedsETB will generate hypotheses, mathematical models, and experiments from the discussion towards further integration of evolutionary ideas towards therapeutic strategies for participants. The pedsETB will collect data through a chart review regarding adherence and results of ETB recommendation.

SUMMARY:
To evaluate the ability of a multidisciplinary and multisite group, the Pediatric Evolutionary Tumor Board (pedsETB), to develop additional therapeutic strategies in patients without curative options or with suboptimal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be considered likely incurable given the standard of care. This is inclusive of patients newly diagnosed, relapsed or in remission but at high risk of recurrence, with suboptimal responses to previous therapy, or with many potentially beneficial, but unlikely curative options for care.

The site investigator will make this determination based on their experience.

* Participant must have an age-appropriate performance status: Karnofsky 50 or more for patients 16 years of age or older OR Lansky score of 50 or more for patients less than16 years of age.
* Participant and/or parents or legal guardian and primary oncologist must be willing to consider the therapeutic strategies recommended by the pedsETB.
* Participant must be willing to be followed over time and allow collection of clinical data including scans, available blood and lab samples, and optional pedsETB serial blood sampling.
* All Participants and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent or assent document.

Exclusion Criteria:

* Participants without known therapies to reliably induce a response are excluded from pedsETB and should seek clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are patients at participating pedsETB sites.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the pedsETB developing therapeutic strategies | Baseline to up to 60 months from end of therapy
  The investigators will measure the ability of a multidisciplinary group, the pedsETB, to develop additional therapeutic strategies in patients without curative options. The investigators plan to enroll 35 patients on the study.
  The primary objective will be successfully met if the pedsETB can develop an evolutionary based therapeutic strategy that differs from the oncologist's opinion prior to presentation for at least 80%, or 28 of these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Metts, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States